CLINICAL TRIAL: NCT00256685
Title: A Double-Blind, Randomized, Placebo-Controlled Efficacy and Safety Study of DVS-233 SR for Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Study Evaluating DVS-233 SR to Treat Vasomotor Systems Associated With Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3151A2-319
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Menopause; Hot Flashes; Sleep Disorders
Keywords: Menopause
MeSH Terms: conditions — Hot Flashes; Sleep Wake Disorders

INTERVENTIONS:
Drug: DVS-233 SR

SUMMARY:
The purpose of this study is to assess the safety and efficacy of desvenlafaxine succinate (DVS) for treatment of moderate to severe vasomotor symptoms (VMS) that are associated with menopause, and also to assess the effects of DVS on sleep parameters and health outcomes indicators.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women who seek treatment for hot flushes
* Minimum of 7 moderate to severe hot flushes per day or 50 per week recorded for 7 consecutive days during screening
* Body Mass Index (BMI) less than or equal to 40 kg/m2

Other inclusions apply.

Exclusion Criteria:

* Hypersensitivity to Venlafaxine
* History of seizure disorder
* History of myocardial infarction or unstable angina within 6 months

Other exclusions apply.

Min Age: 0 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 568
Dates: Start 2004-09; Study Completion 2005-07

PRIMARY OUTCOMES:
Reduction in average daily number of moderate & severe hot flushes and average daily severity score at weeks 4 & 12

SECONDARY OUTCOMES:
Sleep, mood

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer